CLINICAL TRIAL: NCT04914754
Title: Mechanisms Underlying Long-term Fatigue and Exercise Intolerance Following SARS-CoV-2 Infection (COVID-19)
Brief Title: Mechanisms Underlying Long-term Fatigue and Exercise Intolerance Following COVID-19
Acronym: MEXICO
Status: Completed | Type: Observational
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Other Study IDs: 137711
Record Dates: First submitted 2021-04-26; First posted 2021-06-07 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: COVID-19
Keywords: Long COVID; Exercise intolerance; Quality of Life; Coronavirus
MeSH Terms: conditions — COVID-19; Post-Acute COVID-19 Syndrome; Coronavirus Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Whole blood, plasma and serum.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Long COVID with mild exercise impairment: Patients with prior serological or clinical diagnosis of CoV-2 infection and a referred to the UCLH Long-COVID clinic for persistent fatigue or exercise intolerance.
- Healthy Control: Healthy sex-matched and age-matched to within 5 years of Long Covid participants were recruited from UCL staff and students.
- Long COVID with severe exercise impairment: Patients with prior serological or clinical diagnosis of CoV-2 infection and a referred to the UCLH Long-COVID clinic for persistent fatigue or exercise intolerance and an abnormal walk test criteria included: peripheral oxygen desaturation, <85% predicted walk distance, a lactate rise> 1.0 from baseline or a Borg score > 5 for breathlessness or fatigue at end of test.

SUMMARY:
The MEXICO study is an observational study that aims to identify underlying mechanisms contributing to exercise intolerance in the presence of persistent COVID-19 symptoms (Long COVID).

DETAILED DESCRIPTION:
Persistent symptoms of fatigue and severe exercise intolerance have been observed in some patients following infection with CoV-2. Termed 'Long COVID', these symptoms may persist for months after the acute infection has resolved. The mechanisms underlying exercise intolerance in Long COVID are not fully understood and could be the result of dysfunction at any point along the transfer pathway of oxygen from atmosphere to skeletal muscle (uptake in the lungs, heart and blood vessel function and metabolism within skeletal muscle).

The primary objective of the MEXICO study was to identify underlying mechanisms that contributed to exercise intolerance in the presence of persistent covid-19 symptoms (long COVID). Initially it was planned that this would involve a comparison of people with long COVID with and without exercise intolerance. It became clear that recruitment to these two groups was unlikely to complete as while most people with long COVID had some degree of exercise intolerance, severe exercise intolerance was infrequent. Consequently the study was revised to include a reference group of healthy individuals with the primary analysis focusing on a comparison of people with and without long COVID. A comparison of people with long COVID with or without severe exercise intolerance was retained as a secondary exploratory analysis. Ethical approval for the measurements conducted in healthy control subjects was granted by the UCL research ethics Committee.

Revised sample size calculations for study were based on a two-sample t-test (equal variance for simplicity - although the planned analysis would be using a doubly robust potential outcomes method accounting for potential confounders). Sample size estimates were performed using GPower 3.1.9.7 (alpha = 0.05 (two-tailed) and 80% power) assuming that the minimum clinically important difference for the primary outcomes corresponded to a standardized effect size of 0.88 based on previous studies (typically this represents a 10-20% difference in outcome measure). The study was designed to recruit cases and controls in an approximate proportion of 2:1 to enhance the power of the planned substudy analysis. On this basis 32 and 16 participants were required in the long COVID case and healthy group respectively (48 in total).

ELIGIBILITY:
Inclusion Criteria:

* Serological or clinical diagnosis of CoV-2 infection
* Ability to provide written informed consent.

Exclusion Criteria:

* < 18 years old.
* Considered a vulnerable adult
* Participant unwilling to consent
* Terminal illness or severe comorbidities affecting attendance or study investigations
* Pregnancy
* If the participant is not willing to give their consent for a clinical advisor to contact them if necessary
* Inability or presence of a contra-indication for exercise testing
* Chronic oral corticosteroid use (e.g. any maintenance dose of oral steroid, 4 or more course of oral steroid in previous 12 months, but not including prescription of dexamethasone during the acute episode of COVID-19, as long as that has been discontinued).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population (n=51) are either patients with symptoms of Long COVID who have been referred for clinical investigation (with or without severe exercise impairment) or healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2021-05-07 (Actual); Primary Completion 2022-06-20 (Actual); Study Completion 2023-01-17 (Actual)

PRIMARY OUTCOMES:
Pulmonary function (spirometry) | Baseline
  Pulmonary function (ratio of forced expiratory volume in 1 second (FEV1) to forced vital capacity (FVC) (FEV1/FVC)), measured using spirometry, is a co-primary outcome. Compare pulmonary function between long COVID patients with and without severe exercise impairment.
Cardiac function (echocardiography) | Baseline
  Cardiac function (ejection fraction), measured by echocardiography, is a co-primary outcome. Characterise and compare cardiac function between long COVID patients with and without severe exercise impairment.
Microvascular function (microvascular reactivity) | Baseline
  Microvascular reactivity, measured by near-infrared Spectroscopy (NIRS), is a co-primary outcome. Characterise and compare microvascular function between long COVID patients with and without severe exercise impairment.
Macrovascular function (central BP) | Baseline
  Central blood pressure, measured by pulse wave analysis, is a co-primary outcome. Characterise and compare macrovascular function between long COVID patients with and without severe exercise impairment.
Skeletal muscle oxidative capacity | Baseline
  Skeletal muscle oxidative capacity (assessed as the rate of oxygen consumption recovery post-exercise), measured using NIRS, is a co-primary outcome. Characterise and compare skeletal muscle oxidative capacity between long COVID patients with and without severe exercise impairment.

SECONDARY OUTCOMES:
Change in cardiorespiratory fitness (VO2max) | Baseline and 9 months
  Compare changes in VO2max, measured on cardiopulmonary exercise testing, to changes in key markers of the oxygen transport pathway (the primary outcomes).

CONTACTS AND LOCATIONS:
Overall Officials: Professor Hughes, Principal Investigator — UCL, University College London
Locations (1):
- University College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jones S, Tillin T, Williams S, Eastwood SV, Hughes AD, Chaturvedi N. Type 2 diabetes does not account for ethnic differences in exercise capacity or skeletal muscle function in older adults. Diabetologia. 2020 Mar;63(3):624-635. doi: 10.1007/s00125-019-05055-w. Epub 2019 Dec 9. PMID 31820039
- [Background] Jones PW, Beeh KM, Chapman KR, Decramer M, Mahler DA, Wedzicha JA. Minimal clinically important differences in pharmacological trials. Am J Respir Crit Care Med. 2014 Feb 1;189(3):250-5. doi: 10.1164/rccm.201310-1863PP. PMID 24383418
- [Background] Casaburi R. Factors determining constant work rate exercise tolerance in COPD and their role in dictating the minimal clinically important difference in response to interventions. COPD. 2005 Mar;2(1):131-6. doi: 10.1081/copd-200050576. PMID 17136973